CLINICAL TRIAL: NCT06907888
Title: A Confirmatory Study to Evaluate the Rhythm Express Wearable System vs. Simultaneous Polysomnography (PSG) for the Diagnosis of Obstructive Sleep Apnea in an Adult Population With Observed or Suspected Atrial Fibrillation, and Are Indicated for Ambulatory Cardiac Monitoring
Brief Title: Rhythm Express Wearable System vs. Simultaneous Polysomnography for the Diagnosis of Obstructive Sleep Apnea in Adults With Suspected or Observed Atrial Fibrillation
Status: Completed | Type: Observational
Sponsor: VivaQuant (Industry)
Responsible Party: Sponsor
Other Study IDs: VIVA-006
Record Dates: First submitted 2025-03-26; First posted 2025-04-02 (Actual); Last update posted 2025-07-23 (Actual); Status verified 2025-07

CONDITIONS: Obstructive Sleep Apnea (OSA); Atrial Fibrillation (Paroxysmal); Palpitations
Keywords: Obstructive Sleep Apnea; RX-1 mini; Rhythm Express Wearable System; VivaQuant; Atrial Fibrillation
MeSH Terms: conditions — Sleep Apnea, Obstructive; Atrial Fibrillation

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (1):
- Rhythm Express Wearable System: Individuals with suspected or observed paroxysmal atrial fibrillation.
  Interventions: Device: Rhythm Express Wearable System

INTERVENTIONS:
Device: Rhythm Express Wearable System — The Rhythm Express Wearable System consists of the FDA-cleared RX-1 mini Cardiac Monitor, an FDA-cleared pulse oximeter, and a cellular gateway to relay data from the pulse oximeter to the cloud-based RS-1 Server. The RS-1 Sleep Algorithm is a cloud-based software as a medical device (SWMD) that receives inputs from the two FDA-cleared wearable devices. The Algorithm, together with the two wearable devices, comprises the Rhythm Express Wearable System.

SUMMARY:
The goal of this observational study is to confirm the accuracy of the sleep algorithm (software) used in the Rhythm Express Wearable System to detect sleep apnea severity. The study involves participants wearing the RX-1 mini cardiac monitor on their chest and a pulse oximeter during a traditional sleep test, known as polysomnography (PSG), conducted in a sleep center. The performance of the device will be evaluated by comparing the results from the Rhythm Express Wearable System with those from the traditional Polysomnography(PSG).

Participants will:

1. Complete a Screening Visit to confirm they are eligible to participate in the study.
2. Be trained on the use of the Rhythm Express Wearable System.
3. Wear the RX-1 mini cardiac monitor on their chest for 3-5 days/nights.
4. Wear a pulse oximeter for 2 nights before a scheduled sleep study.
5. Complete a sleep study while wearing the Rhythm Express Wearable System.
6. Complete a telephone follow-up visit 5-10 days after the sleep study.

DETAILED DESCRIPTION:
AF is a chronic, progressive, and debilitating cardiovascular disease that exacerbates other cardiovascular diseases and is a leading cause of morbidity (associated illness) and mortality (death). In addition, AF is the most common cardiac arrhythmia that leads to more hospitalizations than any other arrhythmia. Sleep disorders are also associated with a threefold increased mortality and literature suggests a doubled risk for stroke in people with OSA. Identification of OSA and treatment with CPAP is associated with a reduction in the stroke risk for OSA. Thus, early identification and treatment of AF and OSA may be of major societal benefit in reducing mortality and morbidity.

The Rhythm Express Wearable System consists of the RX-1 mini Cardiac Monitor, a Nonin or Viatom Pulse Oximeter, and an Android Cell Phone with the Rhythm Express Oximetry Application. The RS-1 Sleep Algorithm is a cloud-based software as a medical device (SWMD) that receives inputs from the two FDA-cleared wearable devices. The Algorithm, together with the two wearable devices, comprises the Rhythm Express Wearable System.

This multi-center, prospective, observational, confirmatory study is designed to compare sleep apnea severity classification provided by the RS-1 Sleep Algorithm with Polysomnography (PSG). The proposed research will confirm the accuracy of using the Rhythm Express Wearable System to detect apnea/hypopnea index of at least 5/15/30 in patients with observed or suspected atrial fibrillation by comparing it to data recorded in a PSG, which is considered to be the gold standard for sleep testing. In addition, the ability of the RX-1 mini to detect sleep and assess posture and respiratory rate during sleep will be evaluated.

This initiative represents a significant step towards simplifying the screening process for sleep disorders in people indicated for ambulatory cardiac monitoring.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female between 21-85 years of age at the time of informed consent.
2. Subject has a documented or suspected atrial fibrillation.
3. Subject has an indication for 48+ hours of cardiac monitoring due to non-sustained/paroxysmal atrial arrhythmias.
4. STOP-BANG ≥ 2.
5. Subject has capable cellular service at home.
6. Willingness and ability to comply with the study protocol, including informed consent, all study visits, and the collection of adverse events at the telephone follow-up visit.
7. Life expectancy > 6 months.
8. Well-defined and stable diurnal behaviors and nocturnal sleep pattern defined as:

   1. Subject sets aside ample time to sleep to avoid insufficient sleep.
   2. Subject does not do shift work (work outside of the traditional 9 to 5 shift).

Exclusion Criteria:

1. Uses short acting nitrates within 3 hours of the sleep study.
2. Has a permanent pacemaker or ICD.
3. Sustained atrial fibrillation or sustained supraventricular arrhythmias.
4. Known congestive heart failure Class ≥ 1 or known LVEF < 45%.
5. Active acute pulmonary exacerbation (e.g., pneumonia or bronchitis).
6. Known serious respiratory or central nervous system disease that may alter respiratory pattern.
7. Currently participating in or plans to participate in another study that could confound the results of this study.
8. Cognitive or mental health status that would interfere with study participation and/or proper informed consent.
9. Presence of other active medical conditions which could significantly alter pulmonary function.
10. Recent (within 28 days) or expected (during study participation) travel over four or more time zones.
11. History of opioid usage within the past 30 days.
12. Diagnosis of insomnia that is not controlled by medication or other means.
13. Currently using CPAP machine.

Ages: 21 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will include up to 30 adults (21 to 85 years of age, inclusive) with observed or suspected atrial fibrillation who are indicated for ambulatory cardiac monitoring. Enrollment strategies will aim to target the following populations to ensure proper representation of the following underrepresented populations:
  1. Female subjects (N=9-10; ~30%).
  2. Underrepresented minority populations such as African Americans, Asians, Hispanics, etc. (N=6-9; ~20-30%).
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2024-11-18 (Actual); Primary Completion 2025-06-16 (Actual); Study Completion 2025-06-25 (Actual)

PRIMARY OUTCOMES:
Sensitivity and Specificity (AHI>5) | 1 night
  Sensitivity and specificity for detecting an apnea-hypopnea index (AHI) >5, when compared to the adjudicated PSG results.

SECONDARY OUTCOMES:
Sensitivity and Specificity (AHI>15) | 1 night
  Sensitivity and Specificity for detecting an apnea-hypopnea index (AHI) >15, when compared to the adjudicated PSG results.
Body Position | 1 night
  Body position of sleeping subject as measured by the percentage of instances where at least one of the estimated directions in the pair (e.g., LeftSupine) matches the PSG adjudication.

CONTACTS AND LOCATIONS:
Overall Officials: Brian Brockway, Study Director — VivaQuant
Locations (4):
- United States (4):
  - Central Arkansas Lung- J&L Research, Conway, Arkansas
  - Clayton Sleep Institute, St Louis, Missouri
  - Javara - Tryon Medical Partners, PLLC, Charlotte, North Carolina
  - Marshfield Clinic Research Institute, Marshfield, Wisconsin

IPD SHARING:
Plan to Share IPD: Undecided